CLINICAL TRIAL: NCT05302830
Title: Snackability Trial
Brief Title: Effectiveness of the Snackability Smartphone Application to Improve Quality of the Snack Intake, General Diet Quality, and Weight Among College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Principal Investigator, Cristina Palacios, PhD, Associate Professor, Florida International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20-0275
Record Dates: First submitted 2022-03-12; First posted 2022-03-31 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Obesity; Diet, Healthy
MeSH Terms: conditions — Obesity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Snackability app (Experimental): This app allows user to search for a snack (scan barcode or type snack name), add a portion size consumed based on a portion size guide, and then provide a snack score and breakdown scores with a specific feedback message about the score.25 A score ranging from 0-10 points was designed taking into account the first ingredient, the nutrient standard by portion size, and the processing of foods (score ranging from -1 to 1 was subtracted or added depend on processed food classification). The final score ranged from -1 to 11 points. The higher the score, the more compliant it is to the guideline; therefore, the healthier the snack is. The app also provides gamification features as self-motivation (level up and achievement gained) and reporting features as goal-setting and self-monitoring (average daily score and consumed snack history).
  Interventions: Behavioral: Snackability app
- Control group (Placebo Comparator): The control group received a 1-page with information on what is a healthy snack from the USDA: https://www.fns.usda.gov/cn/tools-schools-focusing-smart-snacks. They were given access to the app after the 12-week study period.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Snackability app — This app allows user to search for a snack (scan barcode or type snack name), add a portion size consumed based on a portion size guide, and then provide a snack score and breakdown scores with a specific feedback message about the score.25 A score ranging from 0-10 points was designed taking into account the first ingredient, the nutrient standard by portion size, and the processing of foods (score ranging from -1 to 1 was subtracted or added depend on processed food classification). The final score ranged from -1 to 11 points. The higher the score, the more compliant it is to the guideline; therefore, the healthier the snack is. The app also provides gamification features as self-motivation (level up and achievement gained) and reporting features as goal-setting and self-monitoring (average daily score and consumed snack history).
  Arms: Snackability app
Behavioral: Control group — The control group received a 1-page with information on what is a healthy snack from the USDA: https://www.fns.usda.gov/cn/tools-schools-focusing-smart-snacks. They were given access to the app after the 12-week study period.
  Arms: Control group

SUMMARY:
The Snackability was a two-arm, 12-week randomized control trial among 272 overweight college students. Participants were equally randomized to the intervention group (access to the app) or control group (no access to the app). Diet and weight were assessed at baseline, at 4 weeks, at 8 weeks, and at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese college students-
* Aged 18-24 years
* Owner of a smartphone with Android or iOS platforms with access to an internet connection to use the app
* Willingness to participate in a clinical trial of 3 months and complete assessments at baseline and every 4 weeks at home

Exclusion Criteria:

* Nutrition students
* Enrolled in a weight loss and/or nutrition program
* Taking medications known to influence weight
* Pregnant or breastfeeding

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 272 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Change in general diet quality | 12 weeks
  The change in diet quality was measured using the Healthy Eating Index (HEI) 2015, which was calculated from three 24-h recalls (2 on weekdays and 1 during the weekend) collected at baseline and 12 weeks.
Change in snack quality | 12 weeks
  The change in snacks consumed was recorded from the 24-h recalls collected at baseline and again at 12 months. For each snack consumed at each time point, a score was calculated using the Snackability scoring system.
Change in snack patterns | 12 weeks
  The change in snack patterns was assessed by responses to the survey about intake of snacks completed at baseline and 12 weeks

SECONDARY OUTCOMES:
Change in weight | 12 weeks
  The change in weight was measured between weight measured at baseline and weight measured 12 weeks later

CONTACTS AND LOCATIONS:
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No